CLINICAL TRIAL: NCT00538161
Title: Effect of Low Tidal Volume Ventilation in Improving Oxygenation and Thus Reducing Acute Lung Injury in the Cardiac Surgical Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Sugantha Sundar, Assistant Professor of Anaesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2007P000113
Record Dates: First submitted 2007-09-30; First posted 2007-10-02 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute lung injury; cardiac surgery; The incidence of ARDS after elective cardiac surgery is 1-3%; The impairment of lung function and oxygenation may occur in 20-80% of patients undergoing surgery.; The purpose of this study is to assess the efficacy of low tidal volume ventilation.; Reducing interleukin and cytokine production may prevent or reduce the incidence of acute lung injury.
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low tidal volume arm (Experimental)
  Interventions: Other: Ventilation strategy
- Conventional tidal volume arm (Active Comparator)
  Interventions: Other: Ventilation strategy

INTERVENTIONS:
Other: Ventilation strategy

SUMMARY:
We propose that as low tidal volume ventilation has proven to be beneficial in patients with established ARDS it may have a role in preventing the onset of acute lung injury in the cardiac surgical population. Institution of low tidal volume ventilation in the operating room may reduce the release of the cytokines and interleukins that have been known to contribute to the development of acute lung injury. In this study, we propose that the institution of low tidal volume ventilation in the operating room will reduce the incidence of acute lung injury. Measurement of PaO2 to FiO2 ratio twenty four and forty eight hours post operatively will help determine if there is a difference in oxygenation between the two groups. Chest X-ray findings, time to extubation and length of ICU stay will also determine if there is a role for low tidal volume ventilation in the operating room. We will also attempt to establish a causative mechanism by measuring plasma levels of cytokines known to be associated with the development of ARDS.

DETAILED DESCRIPTION:
Methods- A single center randomized controlled trial was undertaken in 149 patients comparing ventilation with 6 ml/kg TV to ventilation with 10 ml/kg TV in patients undergoing elective cardiac surgery. Study ventilator settings were applied immediately after induction of anesthesia and continued throughout surgery and the subsequent Intensive Care Unit stay. The primary endpoint of the study was time to extubation. Secondary endpoints included the proportion of patients extubated at 6 hours, indices of lung mechanics and gas exchange as well as patient clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients coming in for cardiac surgical procedures will be recruited into the study.
* Both men and women will be recruited into the study.
* All patients over the age of 18 will be recruited into the study.
* Discussion between the surgeon and the primary investigator will happen prior to approaching the patient to obtain informed consent.

Exclusion Criteria:

* Patients with preexisting respiratory failure and active infection will be excluded from the study.
* Patients undergoing one lung ventilation during surgery will be excluded from the study.
* Patients undergoing emergency cardiac surgery will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Time to extubation | the time patient was extubated in the ICU

SECONDARY OUTCOMES:
Oxygenation at 4 hours, 8 hours, 12 hours and 24 hours post surgery. | measurement of blood gas at 4, 8 , 12 and 24 hours post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Talmor, MD, Study Director — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States